CLINICAL TRIAL: NCT01802632
Title: Safety, Tolerability, Pharmacokinetics and Anti-tumour Activity of AZD9291 in Patients With Advanced Non Small Cell Lung Cancer Who Progressed on Prior Therapy With an Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor Agent
Brief Title: AZD9291 First Time In Patients Ascending Dose Study
Acronym: AURA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5160C00001; 2012-004628-39 (EudraCT Number)
Record Dates: First submitted 2013-02-25; First posted 2013-03-01 (Estimated); Results first posted 2016-10-06 (Estimated); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Advanced Non Small Cell Lung Cancer; Advanced (Inoperable) Non Small Cell Lung Cancer
Keywords: Oncology,; Non Small Cell Lung Cancer,; Metastatic,; EGFR sensitivity mutation,; T790M resistance mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Neoplasm Metastasis | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Daily dose of AZD9291 (Experimental): Daily oral dose of AZD9291
  Interventions: Drug: AZD9291

INTERVENTIONS:
Drug: AZD9291 — Starting dose 20 mg, administered once daily. If tolerated subsequent cohorts will test increasing doses of AZD9291, until a maximum tolerated dose or maximum feasible dose is defined

SUMMARY:
This study will treat patients with advanced NSCLC who have already received at least one course of specific anti-cancer treatment but the tumour has started to re-grow following that treatment. This is the first time this drug has ever been tested in patients, and so it will help to understand what type of side effects may occur with the drug treatment, it will measure the levels of drug in the body, it will also measure the anti-cancer activity. By using these pieces of information together the best dose of this drug to use in further clinical trials will be selected.

DETAILED DESCRIPTION:
A Phase I/II, Open-Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Anti-tumour Activity of Ascending Doses of AZD9291 in Patients with Advanced Non Small Cell Lung Cancer who have Progressed Following Prior Therapy with an Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor Agent (AURA)

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analyses
* Aged at least 18 years. Patients from Japan aged at least 20 years.
* Histological or cytological confirmation diagnosis of Non Small Cell Lung Cancer (NSCLC).
* Radiological documentation of disease progression while on a previous continuous treatment with an EGFR TKI e.g. gefitinib or erlotinib (with the exception of 1st line expansion cohort). In addition other lines of therapy may have been given. All patients must have documented radiological progression on the last treatment administered prior to enrolling in the study.
* Patients (with the exception of 1st line expansion cohort) must fulfil one of the following:

  * Confirmation that the tumour harbours an EGFR mutation known to be associated with EGFR TKI sensitivity (including G719X, exon 19 deletion, L858R, L861Q) OR
  * Must have experienced clinical benefit from EGFR TKI, according to the Jackman criteria (Jackman et al 2010) followed by systemic objective progression (RECIST or WHO) while on continuous treatment with EGFR TKI.
* Previous treatment with a single-agent EGFR TKI (e.g. gefitinib or erlotinib).
* Females should be using adequate contraceptive measures, should not be breast feeding and must have a negative pregnancy test prior to start of dosing or evidence of non-child bearing potential.
* Male patients should be willing to use barrier contraception.
* For 1st Line expansion cohort ONLY, confirmation that the tumour is EGFRm+ve and have had no prior therapy for their advanced disease (for 1st line patients biopsy will be at time of diagnosis of advanced disease).
* For dose expansion and extension cohorts, patients must also have confirmation of tumour T790M mutation status (confirmed positive or negative) from a biopsy sample taken after disease progression on the most recent treatment regimen (irrespective of whether this is EGFR TKI or chemotherapy).

Prior to entry a result from the central analysis of the patient's T790M mutation status must be obtained.

- World Health Organisation (WHO) performance status 0-1 with no deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks.

Exclusion Criteria:

* Treatment with an EGFR TKI (erlotinib or gefitinib) within 8 days (approximately 5x half-life) of the first dose of study treatment.
* Any cytotoxic chemotherapy, investigational agents or other anticancer drugs from the treatment of advanced NSCLC from a previous treatment regimen or clinical study within 14 days of the first dose of study treatment.
* AZD9291 in the present study (ie, dosing with AZD9291 previously initiated in this study).
* Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, active bleeding diatheses, or active infection.
* Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 603 (Actual)
Dates: Start 2013-03-04 (Actual); Primary Completion 2015-05-01 (Actual); Study Completion 2023-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuri Rukazenkov, Study Director — AstraZeneca
Locations (39):
- United States (6):
  - Research Site, Aurora, Colorado
  - Research Site, Atlanta, Georgia
  - Research Site, Boston, Massachusetts
  - Research Site, Charlotte, North Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
- Australia (3):
  - Research Site, Heidelberg
  - Research Site, Kogarah
  - Research Site, Nedlands
- France (3):
  - Research Site, Pierre-Bénite
  - Research Site, Saint-Herblain
  - Research Site, Villejuif
- Germany (3):
  - Research Site, Cologne
  - Research Site, Essen
  - Research Site, Würzburg
- Italy (3):
  - Research Site, Genova
  - Research Site, Orbassano
  - Research Site, Roma
- Japan (14):
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Habikino-shi
  - Research Site, Hirakata-shi
  - Research Site, Hiroshima
  - Research Site, Kanazawa
  - Research Site, Kashiwa
  - Research Site, Kobe
  - Research Site, Matsuyama
  - Research Site, Okayama
  - Research Site, Shinjuku-ku
  - Research Site, Sunto-gun
  - Research Site, Takatsuki-shi
  - Research Site, Yokohama
- Research Site, Seoul, South Korea
- Spain (2):
  - Research Site, Madrid
  - Research Site, Seville
- Taiwan (2):
  - Research Site, Tainan
  - Research Site, Taipei
- United Kingdom (2):
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Murat-Onana ML, Ramalingam SS, Janne PA, Gray JE, Ahn MJ, John T, Yatabe Y, Huang X, Rukazenkov Y, Javey M, Brown H, Li-Sucholeiki X. EGFR mutation testing across the osimertinib clinical program. Lung Cancer. 2025 Jun;204:108549. doi: 10.1016/j.lungcan.2025.108549. Epub 2025 Apr 18. PMID 40311309
- [Derived] Martin ML, Correll J, Walding A, Ryden A. How patients being treated for non-small cell lung cancer value treatment benefit despite side effects. Qual Life Res. 2022 Jan;31(1):135-146. doi: 10.1007/s11136-021-02882-6. Epub 2021 May 31. PMID 34056687
- [Derived] Ahn MJ, Han JY, Kim DW, Cho BC, Kang JH, Kim SW, Yang JC, Mitsudomi T, Lee JS. Osimertinib in Patients with T790M-Positive Advanced Non-small Cell Lung Cancer: Korean Subgroup Analysis from Phase II Studies. Cancer Res Treat. 2020 Jan;52(1):284-291. doi: 10.4143/crt.2019.200. Epub 2019 Jul 23. PMID 31345012
- [Derived] Ahn MJ, Tsai CM, Shepherd FA, Bazhenova L, Sequist LV, Hida T, Yang JCH, Ramalingam SS, Mitsudomi T, Janne PA, Mann H, Cantarini M, Goss G. Osimertinib in patients with T790M mutation-positive, advanced non-small cell lung cancer: Long-term follow-up from a pooled analysis of 2 phase 2 studies. Cancer. 2019 Mar 15;125(6):892-901. doi: 10.1002/cncr.31891. Epub 2018 Dec 4. PMID 30512189
- [Derived] Oxnard GR, Hu Y, Mileham KF, Husain H, Costa DB, Tracy P, Feeney N, Sholl LM, Dahlberg SE, Redig AJ, Kwiatkowski DJ, Rabin MS, Paweletz CP, Thress KS, Janne PA. Assessment of Resistance Mechanisms and Clinical Implications in Patients With EGFR T790M-Positive Lung Cancer and Acquired Resistance to Osimertinib. JAMA Oncol. 2018 Nov 1;4(11):1527-1534. doi: 10.1001/jamaoncol.2018.2969. PMID 30073261
- [Derived] Kiura K, Yoh K, Katakami N, Nogami N, Kasahara K, Takahashi T, Okamoto I, Cantarini M, Hodge R, Uchida H. Osimertinib in patients with epidermal growth factor receptor T790M advanced non-small cell lung cancer selected using cytology samples. Cancer Sci. 2018 Apr;109(4):1177-1184. doi: 10.1111/cas.13511. Epub 2018 Feb 27. PMID 29363250
- [Derived] Goss G, Tsai CM, Shepherd FA, Ahn MJ, Bazhenova L, Crino L, de Marinis F, Felip E, Morabito A, Hodge R, Cantarini M, Johnson M, Mitsudomi T, Janne PA, Yang JC. CNS response to osimertinib in patients with T790M-positive advanced NSCLC: pooled data from two phase II trials. Ann Oncol. 2018 Mar 1;29(3):687-693. doi: 10.1093/annonc/mdx820. PMID 29293889
- [Derived] Ramalingam SS, Yang JC, Lee CK, Kurata T, Kim DW, John T, Nogami N, Ohe Y, Mann H, Rukazenkov Y, Ghiorghiu S, Stetson D, Markovets A, Barrett JC, Thress KS, Janne PA. Osimertinib As First-Line Treatment of EGFR Mutation-Positive Advanced Non-Small-Cell Lung Cancer. J Clin Oncol. 2018 Mar 20;36(9):841-849. doi: 10.1200/JCO.2017.74.7576. Epub 2017 Aug 25. PMID 28841389
- [Derived] Thress KS, Jacobs V, Angell HK, Yang JC, Sequist LV, Blackhall F, Su WC, Schuler M, Wolf J, Gold KA, Cantarini M, Barrett JC, Janne PA. Modulation of Biomarker Expression by Osimertinib: Results of the Paired Tumor Biopsy Cohorts of the AURA Phase I Trial. J Thorac Oncol. 2017 Oct;12(10):1588-1594. doi: 10.1016/j.jtho.2017.07.011. Epub 2017 Jul 24. PMID 28751247
- [Derived] Dearden S, Brown H, Jenkins S, Thress KS, Cantarini M, Cole R, Ranson M, Janne PA. EGFR T790M mutation testing within the osimertinib AURA Phase I study. Lung Cancer. 2017 Jul;109:9-13. doi: 10.1016/j.lungcan.2017.04.011. Epub 2017 Apr 19. PMID 28577957
- [Derived] Ballard P, Yates JW, Yang Z, Kim DW, Yang JC, Cantarini M, Pickup K, Jordan A, Hickey M, Grist M, Box M, Johnstrom P, Varnas K, Malmquist J, Thress KS, Janne PA, Cross D. Preclinical Comparison of Osimertinib with Other EGFR-TKIs in EGFR-Mutant NSCLC Brain Metastases Models, and Early Evidence of Clinical Brain Metastases Activity. Clin Cancer Res. 2016 Oct 15;22(20):5130-5140. doi: 10.1158/1078-0432.CCR-16-0399. Epub 2016 Jul 19. PMID 27435396
- [Derived] Oxnard GR, Thress KS, Alden RS, Lawrance R, Paweletz CP, Cantarini M, Yang JC, Barrett JC, Janne PA. Association Between Plasma Genotyping and Outcomes of Treatment With Osimertinib (AZD9291) in Advanced Non-Small-Cell Lung Cancer. J Clin Oncol. 2016 Oct 1;34(28):3375-82. doi: 10.1200/JCO.2016.66.7162. Epub 2016 Jun 27. PMID 27354477
- [Derived] Thress KS, Brant R, Carr TH, Dearden S, Jenkins S, Brown H, Hammett T, Cantarini M, Barrett JC. EGFR mutation detection in ctDNA from NSCLC patient plasma: A cross-platform comparison of leading technologies to support the clinical development of AZD9291. Lung Cancer. 2015 Dec;90(3):509-15. doi: 10.1016/j.lungcan.2015.10.004. Epub 2015 Oct 9. PMID 26494259
- [Derived] Kim TM, Song A, Kim DW, Kim S, Ahn YO, Keam B, Jeon YK, Lee SH, Chung DH, Heo DS. Mechanisms of Acquired Resistance to AZD9291: A Mutation-Selective, Irreversible EGFR Inhibitor. J Thorac Oncol. 2015 Dec;10(12):1736-44. doi: 10.1097/JTO.0000000000000688. PMID 26473643
- [Derived] Yu HA, Tian SK, Drilon AE, Borsu L, Riely GJ, Arcila ME, Ladanyi M. Acquired Resistance of EGFR-Mutant Lung Cancer to a T790M-Specific EGFR Inhibitor: Emergence of a Third Mutation (C797S) in the EGFR Tyrosine Kinase Domain. JAMA Oncol. 2015 Oct;1(7):982-4. doi: 10.1001/jamaoncol.2015.1066. No abstract available. PMID 26181354
- [Derived] Janne PA, Yang JC, Kim DW, Planchard D, Ohe Y, Ramalingam SS, Ahn MJ, Kim SW, Su WC, Horn L, Haggstrom D, Felip E, Kim JH, Frewer P, Cantarini M, Brown KH, Dickinson PA, Ghiorghiu S, Ranson M. AZD9291 in EGFR inhibitor-resistant non-small-cell lung cancer. N Engl J Med. 2015 Apr 30;372(18):1689-99. doi: 10.1056/NEJMoa1411817. PMID 25923549
- See also: D5160C00001AURA_Protocol_for_AZ_ClinTrials_Website — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=492&filename=D5160C00001AURA_Protocol_for_AZ_ClinTrials_Website.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited to different cohorts. Dose escalation cohort of pre-treated patients in 5 dose groups. Dose expansion cohort (pre-treated) in same 5 dose groups. First line patient cohort. 80mg tablet cohort of pre-treated patients. Japan-only cohort (EGFR T790M+ by cytology). Phase II extension cohort in pre-treated EGFR T790M+ patients.
Pre-assignment Details: 603 patients were enrolled and received treatment.
Groups:
- AZD9291 80mg Extension: Phase II dose extension cohort in pre-treated EGFR T790M mutation positive patients in AZD9291 80mg tablet.
- Dose Escalation: Pre-treated patient cohort in doses 20, 40, 80, 160 and 240mg AZD9291 capsule.
- Dose Expansion: Pre-treated EGFR T790M mutation positive (by central testing) patient cohort. Dose groups were expanded to include more patients.
- First Line: Cohort of patients receiving first-line treatment for EGFRm advanced NSCLC, in 80mg and 160mg AZD9291 capsule.
- 80mg Tablet: US-only cohort of pre-treated EGFR patients receiving the tablet formulation of AZD9291 (80 mg).
- Japan Cytology: Japan-only cohort of patients (EGFR T790M mutation status determined from cytology samples) receiving AZD9291 80 mg tablet.
Period: Overall Study
Arm/Group | AZD9291 80mg Extension | Dose Escalation | Dose Expansion | First Line | 80mg Tablet | Japan Cytology
Started | 201 | 31 | 271 | 60 | 12 | 28
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 201 | 31 | 271 | 60 | 12 | 28
Not completed — Death | 28 | 1 | 38 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 4 | 2 | 7 | 3 | 0 | 1
Not completed — Objective Disease Progression | 1 | 12 | 104 | 6 | 4 | 4
Not completed — Ongoing Study at Data Cut-off | 168 | 16 | 115 | 50 | 6 | 22
Not completed — Other (not specified) | 0 | 0 | 7 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD9291 80mg Extension | Dose Escalation | Dose Expansion | First Line | 80mg Tablet | Japan Cytology | Total
Number analyzed (Participants) | 201 | 31 | 271 | 60 | 12 | 28 | 603
Age, Customized [Number; unit: Participants]
  <50 Years | 30 | 3 | 42 | 8 | 3 | 3 | 89
  >=50-<65 Years | 86 | 19 | 142 | 23 | 6 | 13 | 289
  >=65-<75 Years | 64 | 8 | 59 | 22 | 3 | 9 | 165
  >=75 Years | 21 | 1 | 28 | 7 | 0 | 3 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 20 | 167 | 45 | 8 | 21 | 394
  Male | 68 | 11 | 104 | 15 | 4 | 7 | 209
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 114 | 21 | 160 | 43 | 4 | 28 | 370
  Black Or African American | 1 | 0 | 3 | 0 | 1 | 0 | 5
  Missing | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Not Reported | 4 | 4 | 11 | 1 | 0 | 0 | 20
  Other | 4 | 1 | 2 | 1 | 0 | 0 | 8
  White | 76 | 5 | 95 | 14 | 7 | 0 | 197
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) for Dose Expansion Population
Description: Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT: Complete Response (CR): Disappearance of all target and non-target lesions and no new lesions; Partial Response (PR): >= 30% decrease in the sum of diameters of Target Lesions (compared to baseline) and no new lesions. ORR is the percentage of patients with at least 1 visit response of CR or PR (by investigator assessment) that was confirmed at least 4 weeks later, prior to progression or further anti-cancer therapy.
Time Frame: RECIST tumour assessments every 6 weeks from randomisation until objective disease progression, up to approximately 21 months (at time of analysis)
Population: All pre-treated EGFR T790M mutation positive (by central testing) patients who received at least one dose of AZD9291.
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | Dose Expansion
Number analyzed (Participants) | 175
% of participants | 61.7 [54.1 to 68.9]

2. Primary Outcome: Best Objective Response (BOR) for Dose Escalation Population
Description: Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT: Complete Response (CR): Disappearance of all target and non-target lesions and no new lesions; Partial Response (PR): >= 30% decrease in the sum of diameters of Target Lesions (compared to baseline) and no new lesions; Stable disease (SD): Neither sufficient shrinkage to qualify as a response nor sufficient growth to qualify as progression; Progressive Disease (PD): >= 20% increase in the sum of diameters of TLs and an absolute increase in sum of diameters of >=5mm (compared to the previous minimum sum) or progression of NTLs or a new lesion. Not evaluable (NE): TL response is missing and there is no evidence of progression of NTLs and no new lesions. BOR is the best response (by investigator assessment) a patient has achieved where the order of best to worst is CR, PR, SD, PD, NE prior to or at progression and prior to further anti-cancer therapy.
Time Frame: RECIST tumour assessments every 6 weeks from randomisation until objective disease progression, up to approximately 25 months (at time of analysis)
Population: All pre-treated EGFR T790M mutation positive (by central testing) patients who received at least one dose of AZD9291.
Measure: Number; unit: % of participants
Arm/Group | Dose Escalation
Number analyzed (Participants) | 31
% of participants
  Partial Response | 58.1 [54.1 to 68.9]
  Stable disease | 19.4
  Progressive disease | 16.1
  Not evaluable | 6.5

3. Secondary Outcome: Duration of Response (DoR) for Dose Expansion Population
Description: Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT: Complete Response (CR): Disappearance of all target and non-target lesions and no new lesions; Partial Response (PR): >= 30% decrease in the sum of diameters of Target Lesions (compared to baseline) and no new lesions. DoR was defined as the time from the date of first documented response (CR or PR that was subsequently confirmed) until the date of documented progression (PD) or death in the absence of disease progression (by investigator assessment).
Time Frame: as for outcome 1
Population: All pre-treated EGFR T790M mutation positive (by central testing) patients who received at least one dose of AZD9291.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Dose Expansion: Pre-treated EGFR T790M mutation positive (by central testing) population. Dose groups were expanded to include more patients.
Arm/Group | Dose Expansion
Number analyzed (Participants) | 108
months | 11.1 [8.3 to 13.8]

4. Secondary Outcome: Progression-Free Survival (PFS) for Dose Expansion Population
Description: Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT: Progressive Disease (PD): >= 20% increase in the sum of diameters of TLs and an absolute increase in sum of diameters of >=5mm (compared to the previous minimum sum) or progression of NTLs or a new lesion. PFS is the time from date of first dose until the date of PD (by independent central review) or death (by any cause in the absence of progression) regardless of whether the patient withdrew from AZD9291 therapy or received another anti-cancer therapy prior to progression. Patients who had not progressed or died at the time of analysis were censored at the time of the latest date of assessment from their last evaluable RECIST 1.1 assessment.
Time Frame: as for outcome 1
Population: All pre-treated EGFR T790M mutation positive (by central testing) patients who received at least one dose of AZD9291.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Expansion
Number analyzed (Participants) | 175
months | 9.7 [8.3 to 12.5]

5. Primary Outcome: Objective Response Rate (ORR) for Extension Population
Description: Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT: Complete Response (CR): Disappearance of all target and non-target lesions and no new lesions; Partial Response (PR): >= 30% decrease in the sum of diameters of Target Lesions (compared to baseline) and no new lesions. ORR is the percentage of patients with at least 1 visit response of CR or PR (by independent central review) that was confirmed at least 4 weeks later, prior to progression or further anti-cancer therapy.
Time Frame: RECIST tumour assessments every 6 weeks from randomisation until objective disease progression, up to approximately 12 months (at the time of analysis)
Population: All patients in the 80mg AZD9291 extension part of the study (second line or later, EGFR T790M mutation positive by central testing) who received at least one dose of AZD9291 and had measurable disease (by independent central review) at baseline.
Measure: Number (95% Confidence Interval); unit: % of participants
Groups:
- 80mg AZD9291 Extension: Phase II dose extension cohort in pre-treated EGFR T790M mutation positive patients in AZD9291 80mg tablet.
Arm/Group | 80mg AZD9291 Extension
Number analyzed (Participants) | 199
% of participants | 61.3 [54.2 to 68.1]

6. Secondary Outcome: Best Objective Response (BOR) for 80mg AZD9291 Extension Population
Description: as for outcome 2
Time Frame: as for outcome 5
Population: All patients in the 80mg AZD9291 extension part of the study (second line or later, EGFR T790M mutation positive by central testing) who received at least one dose of AZD9291 and had measurable disease (by investigator assessment) at baseline.
Measure: Number; unit: % of participants
Arm/Group | 80mg AZD9291 Extension
Number analyzed (Participants) | 201
% of participants
  Complete Response | 0.5 [54.1 to 68.9]
  Partial response | 70.1
  Stable disease | 22.9
  Progressive disease | 6.0
  Not evaluable | 0.5

ADVERSE EVENTS:
Time Frame: AEs from start of study drug until 28 days post study treatment discontinuation, up to approximately 25 months (at time of analysis).
Description: Different cohorts started at different times and so some cohorts have collected AE data for a shorter length of time, e.g. Extension cohort was the last cohort and follow up is approximately 12 months at time of analysis. Systematic assessment due to regular investigator assessment at study visits.
Arm/Group | AZD9291 80mg Extension | Dose Escalation | Dose Expansion | First Line | 80mg Tablet | Japan Cytology
Serious Adverse Events (participants affected / at risk) | 41/201 | 9/31 | 78/271 | 14/60 | 4/12 | 4/28
Other Adverse Events (participants affected / at risk) | 191/201 | 31/31 | 265/271 | 60/60 | 12/12 | 24/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9291 80mg Extension (N=201) | Dose Escalation (N=31) | Dose Expansion (N=271) | First Line (N=60) | 80mg Tablet (N=12) | Japan Cytology (N=28)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 7 (7) | 3 (3) | 8 (8) | 2 (2) | 0 (0) | 0 (0)
Salmonella sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 2 (2)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 10 (13) | 2 (2) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Corneal erosion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestine ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Mediastinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain injury (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral cyst (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9291 80mg Extension (N=201) | Dose Escalation (N=31) | Dose Expansion (N=271) | First Line (N=60) | 80mg Tablet (N=12) | Japan Cytology (N=28)
Anaemia (Blood and lymphatic system disorders) | 18 (22) | 6 (7) | 36 (49) | 9 (10) | 0 (0) | 5 (5)
Dry eye (Eye disorders) | 12 (14) | 3 (3) | 20 (21) | 7 (7) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 12 (13) | 2 (3) | 19 (26) | 8 (9) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 30 (31) | 3 (4) | 60 (65) | 9 (11) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 93 (147) | 19 (38) | 144 (219) | 41 (62) | 5 (6) | 9 (9)
Dry mouth (Gastrointestinal disorders) | 13 (13) | 1 (1) | 17 (18) | 4 (4) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 34 (45) | 8 (9) | 72 (96) | 15 (18) | 5 (5) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 27 (28) | 8 (14) | 50 (63) | 23 (36) | 1 (1) | 5 (5)
Vomiting (Gastrointestinal disorders) | 23 (31) | 7 (10) | 48 (73) | 9 (13) | 1 (1) | 1 (1)
Asthenia (General disorders) | 19 (34) | 3 (3) | 25 (36) | 2 (2) | 1 (1) | 0 (0)
Fatigue (General disorders) | 24 (27) | 5 (6) | 64 (68) | 15 (16) | 2 (4) | 0 (0)
Oedema peripheral (General disorders) | 15 (17) | 0 (0) | 20 (22) | 2 (3) | 2 (4) | 0 (0)
Pyrexia (General disorders) | 12 (13) | 1 (1) | 27 (28) | 5 (5) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 14 (16) | 6 (10) | 21 (26) | 2 (3) | 1 (1) | 2 (2)
Paronychia (Infections and infestations) | 40 (48) | 8 (11) | 64 (75) | 23 (23) | 2 (3) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 18 (20) | 6 (15) | 27 (29) | 11 (15) | 4 (4) | 2 (2)
Alanine aminotransferase increased (Investigations) | 12 (13) | 3 (3) | 16 (23) | 6 (10) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 14 (18) | 2 (2) | 19 (27) | 7 (11) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 26 (38) | 1 (1) | 24 (31) | 8 (12) | 0 (0) | 3 (4)
White blood cell count decreased (Investigations) | 15 (19) | 3 (4) | 8 (20) | 10 (17) | 0 (0) | 5 (7)
Decreased appetite (Metabolism and nutrition disorders) | 36 (41) | 12 (18) | 69 (80) | 15 (15) | 3 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 (18) | 4 (4) | 26 (33) | 2 (2) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 27 (29) | 3 (6) | 27 (30) | 6 (7) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 (14) | 3 (4) | 24 (27) | 8 (8) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 15 (16) | 2 (2) | 20 (20) | 0 (0) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 22 (22) | 4 (7) | 30 (34) | 5 (8) | 1 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 19 (21) | 1 (1) | 27 (28) | 7 (10) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 32 (36) | 4 (4) | 55 (64) | 9 (11) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 (19) | 2 (3) | 37 (43) | 2 (2) | 4 (5) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 12 (13) | 3 (3) | 32 (39) | 16 (17) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 43 (45) | 8 (8) | 62 (73) | 24 (29) | 4 (4) | 8 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 25 (29) | 8 (9) | 56 (61) | 14 (15) | 3 (4) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 49 (58) | 11 (17) | 75 (101) | 20 (25) | 2 (2) | 3 (3)
Skin fissures (Skin and subcutaneous tissue disorders) | 12 (12) | 4 (4) | 30 (31) | 9 (9) | 1 (1) | 1 (2)
Leukopenia (Blood and lymphatic system disorders) | 9 (9) | 1 (1) | 10 (16) | 4 (6) | 0 (0) | 3 (6)
Lymphopenia (Blood and lymphatic system disorders) | 5 (5) | 1 (1) | 6 (8) | 1 (1) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 7 (7) | 4 (8) | 12 (12) | 3 (5) | 0 (0) | 4 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (10) | 2 (2) | 20 (25) | 7 (9) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 10 (10) | 3 (3) | 25 (27) | 4 (4) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 8 (8) | 4 (4) | 16 (18) | 4 (4) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (5) | 0 (0) | 11 (11) | 5 (5) | 2 (2) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 3 (3) | 0 (0) | 4 (4) | 8 (10) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 3 (3) | 0 (0) | 8 (10) | 5 (5) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 16 (17) | 7 (7) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 6 (6) | 1 (1) | 5 (6) | 8 (8) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 3 (3) | 1 (1) | 14 (15) | 3 (3) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Pharyngitis (Infections and infestations) | 7 (7) | 0 (0) | 7 (7) | 1 (1) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 10 (10) | 1 (1) | 19 (26) | 2 (3) | 1 (2) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 6 (6) | 0 (0) | 9 (10) | 5 (5) | 1 (1) | 3 (3)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 7 (8) | 3 (3) | 0 (0) | 2 (6)
Neutrophil count decreased (Investigations) | 10 (10) | 3 (6) | 16 (38) | 5 (5) | 0 (0) | 6 (8)
Weight decreased (Investigations) | 6 (6) | 2 (2) | 19 (19) | 13 (13) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 8 (10) | 1 (1) | 1 (3) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 0 (0) | 19 (20) | 6 (6) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 1 (1) | 13 (13) | 4 (4) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (10) | 0 (0) | 19 (22) | 2 (2) | 4 (7) | 0 (0)
Dizziness (Nervous system disorders) | 9 (9) | 1 (1) | 25 (29) | 5 (5) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 4 (4) | 3 (3) | 15 (16) | 10 (12) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1) | 13 (14) | 9 (11) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 0 (0) | 6 (6) | 4 (4) | 1 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 20 (20) | 3 (4) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 11 (12) | 4 (4) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0) | 10 (11) | 6 (6) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 4 (4) | 4 (4) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1) | 9 (9) | 1 (1) | 0 (0) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 (9) | 1 (4) | 11 (15) | 5 (6) | 1 (2) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 14 (15) | 3 (3) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 1 (1) | 7 (8) | 4 (5) | 2 (2) | 0 (0)
Blepharitis (Eye disorders) | 2 (2) | 2 (2) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 4 (4) | 2 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 7 (7) | 2 (2) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 5 (5) | 1 (4) | 4 (4) | 1 (1) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 13 (13) | 3 (3) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 5 (5) | 0 (0) | 4 (4) | 1 (1) | 2 (3) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 1 (1) | 7 (7) | 0 (0) | 2 (4) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Renal function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 7 (7) | 2 (2) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 6 (6) | 3 (3) | 8 (8) | 3 (3) | 0 (0) | 0 (0)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 3 (3) | 7 (7) | 3 (3) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 2 (2) | 7 (7) | 2 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (4) | 0 (0) | 11 (11) | 1 (1) | 2 (2) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 13 (13) | 0 (0) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 11 (11) | 3 (3) | 3 (3) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (4) | 17 (17) | 4 (4) | 1 (1) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 10 (10) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 4 (4) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
All 6 cohorts are still on-going. Data cut-off on 1st May 2015 was for primary analyses in main cohorts of dose escalation, dose expansion, extension. AEs presented for all cohorts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review, should the submission for publication be delayed in order to file patent application. The sponsor cannot require changes to the communication and cannot extend the embargo.